CLINICAL TRIAL: NCT04547933
Title: Correlation Analysis of Quality of Life With Different Groups of Female Lower Urinary Tract Symptoms Based on Bladder Diary
Brief Title: Female LUTS and Quality of Life
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202006086RIND
Record Dates: First submitted 2020-09-08; First posted 2020-09-14 (Actual); Last update posted 2020-09-14 (Actual); Status verified 2020-07

CONDITIONS: Bladder Diary
Keywords: Lower urinary tract symptoms; Quality of life
MeSH Terms: conditions — Lower Urinary Tract Symptoms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- OAB-wet: The bladder diaries and the King's Health Questionnaires of all consecutive women with lower urinary tract symptoms who visited urogynecologic clinics in a tertiary referral center, were reviewed. Based on bladder diaries, women with at least one episode of urgency and urinary incontinence (UI) were allocated to the overactive bladder syndrome (OAB) -wet group.
  Interventions: Diagnostic Test: Bladder diary
- OAB-dry: The bladder diaries and the King's Health Questionnaires of all consecutive women with lower urinary tract symptoms who visited urogynecologic clinics in a tertiary referral center, were reviewed. Based on bladder diaries, women with at least one episode of urgency but without incontinence were allocated to the OAB-dry group.
  Interventions: Diagnostic Test: Bladder diary
- UI: The bladder diaries and the King's Health Questionnaires of all consecutive women with lower urinary tract symptoms who visited urogynecologic clinics in a tertiary referral center, were reviewed. Based on bladder diaries, women with at least one episode of UI but without urgency were allocated to the UI group.
  Interventions: Diagnostic Test: Bladder diary
- Nocturia: The bladder diaries and the King's Health Questionnaires of all consecutive women with lower urinary tract symptoms who visited urogynecologic clinics in a tertiary referral center, were reviewed. Based on bladder diaries, women with more or equal to 2 episodes of nocturia but without urgency and UI were allocated to the nocturia group.
  Interventions: Diagnostic Test: Bladder diary
- Frequency: The bladder diaries and the King's Health Questionnaires of all consecutive women with lower urinary tract symptoms who visited urogynecologic clinics in a tertiary referral center, were reviewed. Based on bladder diaries, women with more or equal to 8 episodes of daytime frequency but without urgency, UI and nocturia were allocated to the frequency group.
  Interventions: Diagnostic Test: Bladder diary
- Normal: The bladder diaries and the King's Health Questionnaires of all consecutive women with lower urinary tract symptoms who visited urogynecologic clinics in a tertiary referral center, were reviewed. Based on bladder diaries, women without urgency, UI, nocturia nor frequency were allocated to the normal group.
  Interventions: Diagnostic Test: Bladder diary

INTERVENTIONS:
Diagnostic Test: Bladder diary — A 3-day bladder diary recording daily drinking fluid amount, daily urine amount, urgency and urinary incontinence episodes.

SUMMARY:
Storage symptoms include frequency, urgency, nocturia and incontinence. Based on bladder diaries, we could get the objective data of the above symptoms. To the best of our knowledge, there is lack of correlation of quality of life with lower urinary tract symptoms based on bladder diaries. Thus, we aimed to perform the study.

DETAILED DESCRIPTION:
The bladder diaries and the King's Health Questionnaires of all consecutive women with lower urinary tract symptoms who visited urogynecologic clinics in a tertiary referral center, were reviewed. Based on bladder diaries, women with at least one episode of urgency and urinary incontinence (UI) were allocated to the overactive bladder syndrome (OAB) -wet group. Women with at least one episode of urgency but without incontinence were allocated to the OAB-dry group. Women with at least one episode of UI but without urgency were allocated to the UI group. Women with more or equal to 2 episodes of nocturia but without urgency and UI were allocated to the nocturia group. Women with more or equal to 8 episodes of daytime frequency but without urgency, UI and nocturia were allocated to the frequency group. Otherwise, normal group. Analysis of variance with Bonferroni correction was used to perform statistical analysis for between-group comparisons.

ELIGIBILITY:
Inclusion Criteria:

* Women with lower urinary tract symptoms
* Finish 3-day bladder diary
* Finish King's Health Questionnaire

Exclusion Criteria:

* Incomplete data
* Pregnant women
* Urinary tract infection, acute or chronic
* History of pelvic malignancy

Ages: 20 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women with lower urinary tract symptoms completed a 3-day bladder diary and King's Health Questionnaire.
Sampling Method: Non-Probability Sample
Enrollment: 2953 (Actual)
Dates: Start 2010-01-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Finish quality of life accessment | January 2010 to December 2019
  Quality of life was accessed by King's Health Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Ho-Hsiung Lin, PhD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No
IPD will be shared under reasonable request

REFERENCES:
- [Result] Haylen BT, de Ridder D, Freeman RM, Swift SE, Berghmans B, Lee J, Monga A, Petri E, Rizk DE, Sand PK, Schaer GN; International Urogynecological Association; International Continence Society. An International Urogynecological Association (IUGA)/International Continence Society (ICS) joint report on the terminology for female pelvic floor dysfunction. Neurourol Urodyn. 2010;29(1):4-20. doi: 10.1002/nau.20798. PMID 19941278
- [Result] Coyne KS, Wein AJ, Tubaro A, Sexton CC, Thompson CL, Kopp ZS, Aiyer LP. The burden of lower urinary tract symptoms: evaluating the effect of LUTS on health-related quality of life, anxiety and depression: EpiLUTS. BJU Int. 2009 Apr;103 Suppl 3:4-11. doi: 10.1111/j.1464-410X.2009.08371.x. PMID 19302497
- [Result] Hsiao SM, Lin HH. Medical treatment of female overactive bladder syndrome and treatment-related effects. J Formos Med Assoc. 2018 Oct;117(10):871-878. doi: 10.1016/j.jfma.2018.01.011. Epub 2018 Feb 15. PMID 29398096
- [Result] Hsiao SM, Su TC, Chen CH, Chang TC, Lin HH. Autonomic dysfunction and arterial stiffness in female overactive bladder patients and antimuscarinics related effects. Maturitas. 2014 Sep;79(1):65-9. doi: 10.1016/j.maturitas.2014.06.001. Epub 2014 Jun 20. PMID 25022469
- [Result] Hsiao SM, Liao SC, Chen CH, Chang TC, Lin HH. Psychometric assessment of female overactive bladder syndrome and antimuscarinics-related effects. Maturitas. 2014 Dec;79(4):428-34. doi: 10.1016/j.maturitas.2014.08.009. Epub 2014 Sep 3. PMID 25238744